CLINICAL TRIAL: NCT05739370
Title: Internet Delivered Psychotherapy for Older Adults: Development and Evaluation of an Online Problem-Solving Therapy Program for Depression.
Brief Title: Internet Delivered Psychotherapy for Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: Hotchkiss Brain Institute, University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB21-1012
Record Dates: First submitted 2023-01-09; First posted 2023-02-22 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-01

CONDITIONS: Depression in Old Age; Depression, Anxiety
Keywords: Online Psychotherapy
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Aging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ger-iPST (Experimental): Prospective participants will be contacted by telephone to confirm eligibility, explain the study protocol, and obtain informed consent. An in-person or videoconference assessment will be used to administer baseline PHQ-9 to confirm enrolment criteria and will be asked questionnaire to gather demographic information. Participants will then be provided with an email link to access the Online Psycho Therapy Tool (OPTT). PHQ-9 will be collected again at the mid-point (4 weeks) and after completing the program through OPTT. Caregivers will be invited to assist the participant if required in completing Ger-iPST modules, and weekly telephone support calls by a research assistant will be provided to assist with any difficulty navigating technical aspects of the Ger-iPST platform.
  Interventions: Other: Problem-Solving Therapy for Older Adults

INTERVENTIONS:
Other: Problem-Solving Therapy for Older Adults — Problem-Solving Therapy for Older Adults (Ger-iPST) is an 8-week online psychotherapy program with online therapist support delivered through the Online Psycho Therapy Tool (OPTT). Ger-iPST has several evidence-based elements tailored to the specific needs of older adults, including relevant content (e.g. aging-related examples); process adaptations (e.g. more repetition); and digital usability modifications (e.g. high-contrast text).
  Ger-iPST contains therapy modules assigned weekly and accessible at any time during the week. Modules begin with a brief, guided mindfulness relaxation exercise, followed by approximately 20 slides taking, on an average 1 hour to complete. Each module highlights a different step of Psychotherapy (PST) and includes an overview of a new skill, interactive activities and examples. A homework exercise designed to guide participants in applying a new PST skill exercise is submitted through the platform, and a clinician will provide personalized feedback.
  Other Names: Ger-iPST

SUMMARY:
The goal of this mixed-methods, single-arm intervention study is to develop and evaluate a new internet-delivered psychotherapy option called Ger-iPST in older adults with symptoms of depression.

The overall aim of this project is to improve access to psychotherapy for older adults by developing, adapting and implementing a new internet-based treatment option, Ger-iPST. Towards this aim, our objectives are to:

1. Examine the preliminary effectiveness of Ger-iPST for symptoms of depression.
2. Examine barriers and facilitators to the use of Ger-iPST.

Participants will be asked to complete 8 weekly online therapy modules (Ger-iPST) through the Online Psycho Therapy Tool (OPTT); each module takes 45-60 minutes, and an extra 20-30 on weekly homework. Caregivers will be invited to assist participants if required.

Homework exercises are submitted through the platform, and a clinician trained in PST l will provide personalized, asynchronous online feedback. Participants will receive a weekly phone call from a research assistant to support any technical issues with completing the online modules. Following completion of the Ger-iPST modules, participants will be interviewed to provide feedback on acceptability and barriers and facilitators to the use of Ger-iPST.

DETAILED DESCRIPTION:
Background & Rationale: Many older adults in the community experience symptoms of depression, but few receive adequate treatment, which can include medications or psychotherapy (talk therapy). Problem-Solving Therapy (PST) is a very effective psychotherapy for depression, but psychotherapy such as PST is usually not available to older adults due to high cost, limited resources, and other barriers such as lack of transportation. Internet-delivered psychotherapy is a more accessible option that can be as effective as traditional face-to-face therapy.

Research Question and Objectives: The overall aim of this project is to improve access to psychotherapy for older adults by developing, adapting and implementing a new evidence-based treatment option, Ger-iPST. Towards this aim, our objectives are to:

1. Develop the Ger-iPST intervention.
2. Examine the effectiveness and implementation of Ger-iPST: 2a. Measure the preliminary effectiveness of symptoms of depression in older adults; 2b. Explore barriers and facilitators to the use of Ger-iPST among participants and experiences with implementation.

Methods: The investigator will implement and evaluate the effectiveness of Ger-iPST in Calgary, Alberta. Ger-iPST is an 8-week online psychotherapy program with online therapist support based on Problem Solving Therapy (PST), a proven and safe psychotherapy for depression in older adults. Ger-iPST will be tailored to the specific needs of older adults with relevant content (e.g. modules using aging-related examples); process adaptations (e.g. more repetition); and digital usability modifications. Participants will complete weekly online Ger-iPST modules, and the investigator will measure symptoms of depression before, during, and after completing the program. The investigator will also collect information on symptoms of anxiety, quality of life, and disability. The Ger-iPST intervention will be hosted on an existing, secure, cloud-based psychotherapy platform, Online PsychoTherapy Tool (OPTT). All quantitative data collection will occur using questionnaires on the platform. Following completion of the Ger-iPST modules, participants will be interviewed to provide feedback on acceptability and barriers and facilitators to the use of Ger-iPST. These results will be used to improve and adapt the resource to best suit the needs of older adults.

Treating depression improves functioning, emotional well-being, and overall health among older adults. Many older adults prefer psychotherapy over (or in addition to) medication for the treatment of depression, and given that a growing number of older adults use the internet, internet-delivered therapy has the potential to greatly improve access to treatment for older adults with depression.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are 65 years or older
* Presenting with a primary complaint of depression and a Patient Health Questionnaire (PHQ)-9 score > 5
* English Speaking
* Residents of Alberta
* Have internet access

Exclusion Criteria:

* Individuals with acute safety concerns (e.g.suicidal ideation), psychotic symptoms, moderate cognitive impairment (Montreal Cognitive Assessment(MoCA) < 21) or currently receiving psychotherapy

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Measure the effectiveness for symptoms of depression in older adults. | Baseline, mid-point (4-weeks) and after completing the program (8-weeks).
  The outcome measures the change in depressive symptoms based on the PHQ-9 score,The 9-items on the PHQ-9 reflect DSM-V diagnostic criteria and are rated from 0 (''not at all") to 3 ("nearly every day") based on self-reported symptoms in the preceding 2-weeks. Scores >5, 10, and 15 indicate mild, moderate, and severe depression symptoms, respectively. The PHQ-9 has been validated for use with older adults in primary care and those with chronic medical illnesses, is relatively brief, and is responsive to change.

SECONDARY OUTCOMES:
Examine implementation outcomes - Anxiety symptoms. | 8 weeks via OPTT.
  • Anxiety symptoms based on the Geriatric Anxiety Inventory (GAI), a 20-item scale developed specifically for measuring anxiety in older adults
Examine implementation outcomes - Disability Assessment. | 8 weeks via OPTT.
  • Disability using the 12-item World Health Organization Disability Assessment Schedule (WHODAS 2.0). The WHODAS measures disability (irrespective of underlying disease) within 6 functional domains: cognition, mobility, self-care, getting along, life activities and participation. Each item is rated on a scale of 0-4; higher scores indicate greater disability
Examine implementation outcomes - Quality of life. | 8 weeks via OPTT.
  • Quality of life using the 34-item Quality of Life in Depression Scale (QLDS). The scale has both positive and negative items; lower scores indicate higher quality of life
Examine implementation outcomes - Usability. | 8 weeks via OPTT.
  • Usability of Ger-iPST will be measured using the 10-item System Usability Scale (SUS) used often and validated in the assessment of the usability of technological interfaces. Items are rated from 0-6 based on the extent to an agreement with statements about ease of use of the software, such as "I felt very confident using the system." Scores are converted to a percentile ranking; higher scores indicate above average usability
Explore barriers and facilitators experienced with implementation. | 8 weeks
  The investigator will use a semi structured interview conducted by telephone or videoconferencing with participants in their own homes. The investigator is doing interviews not focus groups, to maintain the anonymity of participants in the Ger-iPST intervention. We will explore the user experience of Ger-iPST implementation, focusing on the acceptability and usability of the intervention and any barriers or facilitators of implementation. The analysis will be facilitated with NVIVO software.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Kirkham, MD, Principal Investigator — University of Calgary
Locations (1):
- Department of Psychiatry, Cumming School of Medicine, University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No